CLINICAL TRIAL: NCT04455711
Title: The Efficacy of Intravenous Lidocaine With Continuous Infusion of Remifentanil for Attenuating Double Lumen Tube Induced Cough During Emergence
Brief Title: The Effect of Lidocaine on Smooth Emergence With Double Lumen Tube
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiyoung Yoo, Assistant professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AJIRB-MED-OBS-16-342
Record Dates: First submitted 2020-05-06; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Cough; Lidocaine
MeSH Terms: conditions — Cough | interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remifentanil group (Placebo Comparator): Emerge with continuous infusion of remifentanil 1.5 ng/ml
  Interventions: Drug: Remifentanil
- Lidocaine group (Experimental): Emerge with continuous infusion of remifentanil 1.5 ng/ml with IV bolus of lidocaine 1.5 mg/kg
  Interventions: Drug: Lidocaine Iv; Drug: Remifentanil

INTERVENTIONS:
Drug: Lidocaine Iv — Bolus dose of 1.5 mg/kg lidocaine was injected immediate after operation.
  Arms: Lidocaine group
Drug: Remifentanil — Continuous infusion of remifentanil 1.5 ng/ml until extubation

SUMMARY:
Cough suppression during emergence and tracheal extubation from general anaesthesia has become an important issue as part of patient safety. Cough arised from the mechanical irritation of endotracheal tube and cuff could be accompanied by various adverse effects such as laryngospasm, hypertension, tachycardia, arrhythmia and increase of intracranial, intraocular, or intra-abdominal pressure.

Several cough-preventing strategies have been proposed for smooth emergence, such as opioids, dexmedetomidine or lidocaine. Maintenance of remifentanil infusion during emergence has been reported to be an effective method in reducing cough and cardiovascular change without delay of recovery. In previous studies, the effetive effect-site concentraions for 95% of adults (EC95) for preventing cough are a little different depending on anaestheic agent, type of surgery and sex, ranged from 2.14 to 2.94 ng/ml. However, since most of these studies are for sing lumen endotracheal tube, similar preventing effect would not be expected for double lumen tube (DLT) because of its large diameter and long length. Another problem is higher concentration of remifentanil more than 2.5 ng/ml could not guarantee the safety after extubation. The efficacy of a single IV bolus of lidocaine for the prevention of cough has been the subject of numerous trials.

Therefore, combined use of lidocaine and remifentanil could effectively prevent emergence cough for DLT without the risk of high concentration of remifentanil.

ELIGIBILITY:
Inclusion Criteria:

* Patients needs for double lumen tube intubation for one lung ventilation during surgery with ASA (American society of Anesthesiologists) class I or II

Exclusion Criteria:

* Gastroesophageal reflux disease
* Obese patients (BMI > 30)
* Recent upper respiratory infection history (within 3 weeks)
* Asthma history
* Anticipating difficult airway

Ages: 19 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Cough incidence | from the time of end of the operation up to 10 min after extubation

SECONDARY OUTCOMES:
Cough severity | from the time of end of the operation up to 10 min after extubation
  cough severity is graded as follows; mild cough (1 cough without lifting head), moderate cough ( more than 1 cough not sustained more than 5 seconds), severe cough (cough sustained more than 5 seconds)
hoarseness | 30 min at the recovery room

CONTACTS AND LOCATIONS:
Overall Officials: Ji young Yoo, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou University Hospital, Suwon, Gyeonggido, South Korea

IPD SHARING:
Plan to Share IPD: No